CLINICAL TRIAL: NCT05933447
Title: A Randomized, Double-Blind and Nested Crossover (For Placebo and Moxifloxacin) Thorough QT Study to Evaluate the Effect of Rodatristat Ethyl, Rodatristat, and Its Major Metabolites on Cardiac Repolarization in Healthy Volunteers
Brief Title: Thorough QT Study to Evaluate the Effect of Rodatristat Ethyl, Rodatristat and Its Major Metabolites on the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altavant Sciences GmbH (Industry)
Collaborators: Altasciences Clinical Kansas, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RVT-1201-1004
Record Dates: First submitted 2023-05-03; First posted 2023-07-06 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — rodatristat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rodatristat Ethyl (Experimental)
  Interventions: Drug: Rodatristat Ethyl
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Placebo for Rodatristat (Placebo Comparator)
  Interventions: Drug: Placebo for Rodatristat
- Placebo for Moxifloxacin (Placebo Comparator)
  Interventions: Drug: Placebo for Moxifloxacin

INTERVENTIONS:
Drug: Rodatristat Ethyl — Oral, Tablet, 300 mg QD, 300 mg BID, 600 mg BID, 900 mg BID, 900 mg QD
  Arms: Rodatristat Ethyl
Drug: Moxifloxacin — Oral, Tablet, 400 mg QD
  Arms: Moxifloxacin
Drug: Placebo for Rodatristat — Oral, Tablet, O mg QD, 0 mg BID
  Arms: Placebo for Rodatristat
Drug: Placebo for Moxifloxacin — Oral, Tablet, 0 mg QD
  Arms: Placebo for Moxifloxacin

SUMMARY:
To evaluate whether Rodatristat Ethyl prolongs the QTc interval when orally administered to healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase I, single-center, double blind, randomized, placebo- and positive-control, nested crossover study in approximately 64 healthy volunteers. This thorough QT/QTc study will be conducted to evaluate the effect of Rodatristat Ethyl on QT prolongation.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent and to comply with the requirements of the study for its duration.
2. Healthy adult males or females aged 18 to 55 years, inclusive. As determined by the Investigator, healthy subjects are defined as individuals free from clinically significant illness or disease as determined by their medical history, physical examination, vital signs, cardiac monitoring, and clinical laboratory test results.
3. A male subject is eligible to participate if he does not have a female partner who is pregnant or who intends to become pregnant during the study. Male subjects must agree to use contraception.
4. Female subjects of childbearing potential must agree to use contraception.
5. Body mass index (BMI) within 18.0 kg/m2 to 33.0 kg/m2, inclusively.

Exclusion Criteria:

1. Female who is lactating.
2. Positive pregnancy test at the Screening visit or check-in or planning to become pregnant within the next 6 months.
3. Pulse rate less than 40 beats per minute (bpm) or more than 100 bpm at the Screening visit or check-in.
4. A sustained supine systolic blood pressure > 140 mm Hg or < 90 mmHg or a supine diastolic blood pressure > 90 mmHg or < 50 mmHg at the Screening visit, check-in, or prior to dosing.
5. History of significant hypersensitivity to rodatristat ethyl, moxifloxacin, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
6. As determined by the Investigator, any known pre-existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings including, but not limited to a history of clinically significant gastrointestinal (including cholecystectomy), hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, endocrine, immunologic, dermatologic or cardiovascular disease, including:

   1. History of Gilbert's Syndrome
   2. History of depression
   3. History of any allergy that, in the opinion of the Investigator, contraindicates participation in the trial
7. An uninterpretable or abnormal Screening ECG indicating a second or third degree atrioventricular block, presence of out-of-range cardiac interval (heart rate [HR] < 40 bpm, PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and Fridericia-corrected QT interval (QTcF) > 450 msec for males and > 470 msec for females) on the ECG at the Screening visit or other clinically significant ECG abnormalities, unless deemed non significant by an investigator.
8. History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia. Subjects will also be excluded if there is a family history of long QT syndrome or Brugada syndrome.
9. Clinically significant abnormalities in laboratory test results, as determined by the Investigator, (including hepatic and renal panels, complete blood count, coagulation, chemistry panel, and urinalysis) at the Screening visit or check-in that are confirmed by a repeat reading .

   1. Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
   2. Estimated glomerular filtration rate < 80 mL/min/1.73 m2 at the Screening visit, calculated using the Cockcroft-Gault formula
   3. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) values greater than upper limit of normal (ULN). A single repeat measurement is allowed for eligibility determination
   4. Positive urine test for drugs of abuse at the Screening visit or check-in
   5. Positive alcohol test (breath) at the Screening visit or check-in
   6. Positive pregnancy test at the Screening visit or check-in
10. Presence of unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia.
11. Subjects with a clinical history of or current alcohol abuse defined as an average weekly intake of more than 21 units for males or 15 units for females (1 unit = 11 oz beer, 4 oz wine, or 1 oz spirits).
12. Subjects with a clinical history of or current illicit drug use which, in the opinion of the Investigator, would interfere with the subjects ability to complete the study and could compromise subject safety and/or the results of the study.
13. Any clinically significant illness, including viral syndromes, in the 28 days prior to dosing.
14. Use of prescription or nonprescription drugs, (with exception of contraceptive and acetaminophen allowed), including high-dose vitamins, dietary supplements (including St. John's Wort) within 14 days or 5 half-lives of the prescription or nonprescription drug (whichever is longer) prior to the first dose of study drug, through to the final Follow-up visit, unless in the opinion of the Investigator and Sponsor, the medication would not interfere with the study outcomes or compromise subject safety.
15. Consumption of grapefruit and/or pomelo and Seville oranges or their juices within the 7 days prior to dosing and until collection of the final lab sample.
16. Use of medications associated with QT prolongation within 30 days prior to dosing and during the study.
17. Any other clinically significant abnormalities in laboratory test results at the Screening visit or check-in, or any other medical, psychological, or social condition that that would, in the opinion of an investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
18. Previous intake of rodatristat ethyl in the last 6 months before Day 1.
19. Participation in another investigational drug, vaccine, or device study or treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, before dosing, or 90 days for a biologic.
20. Donation of plasma within 7 days prior to dosing or donation or loss of blood (excluding volume drawn at the Screening visit) of 50 mL to 499 mL of blood within 30 days or more than 499 mL within 56 days prior to dosing.
21. Is an employee of the Investigator or study center with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member of the employee or Investigator.
22. Subjects who have smoked or used tobacco or nicotine containing products within 3 months prior to the Screening visit and who are unwilling to refrain from smoking, tobacco use, or use of nicotine products for the entire duration of the study (through the Follow-up visit).
23. Subjects unable to abstain from caffeine, xanthine, or strenuous exercise for 72 hours prior to dosing until collection of the final lab sample.
24. Showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C SSRS) administered at the Screening visit or prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of rodatristat ethyl, rodatristat, and its major metabolites on the Fredericia-corrected QT interval in healthy volunteers using concentration-QT analyses following administration of multiple doses of rodatristat ethyl | 20 Days
  Measure change in baseline in QTcF

SECONDARY OUTCOMES:
Evaluate the effect of multiple doses of rodatristat ethyl on other electrocardiogram (ECG) parameters | 55 Days
  Measure change from baseline in heart rate
Evaluate the pharmacokinetics (PK) of rodatristat ethyl, rodatristat and it's major metabolites following multiple doses of rodatristat ethyl | 55 Days
  Measure PK parameters time to maximum concentration (tmax)
Evaluate effect of multiple doses of rodatristat ethyl on plasma 5-hydroxyindoleacetic acid (5-HIAA) | 55 Days
  Measure change from baseline in plasma 5-HIAA concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No